CLINICAL TRIAL: NCT01082432
Title: Superimposed Electrical Stimulation Real-time Effects on Repeated Muscle Contractions Enable to Increase Recovery From Thumb Joint Stiffness After Surgery of the Ulnar Collateral Ligament
Brief Title: Electrical Stimulation to Recover Greater Range of Motion After Surgery
Status: Completed | Type: Observational
Sponsor: Université Joseph Fourier (Other)
Responsible Party: Université Joseph Fourier - TIMC IMAG laboratory
Other Study IDs: SES 327
Record Dates: First submitted 2010-03-01; First posted 2010-03-08 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-02

CONDITIONS: Thumb Joint Stiffness
Keywords: thumb; Ulnar collateral ligament; superimposed electrical stimulation; stiffness; adhesions
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: electrically induced muscle activation — 30 Hz frequency, 200 µs pulse duration, and 40% duty cycle (4 sec on, 6 sec off)

SUMMARY:
Background

One of the potentially debilitative complications of operative repair and subsequent immobilization is stiffness that appears secondary to inflammation and adhesions. To prevent such a physical impairment, active joint mobilization has shown to be efficient. However, adhesions sometimes remain despite the therapy. Due to the viscoelastic nature of the biological tissues, if a technique can enable to extend the muscle ability to impose a maximal steady stress on adhesions, adhesion deformation should be greater and range of motion deficit should be reduced. Within that context, the purpose of the present study was to assess the real-time effects of superimposed electrical stimulation (SES) on maximal voluntary muscular contraction (VOL) over time and to assess SES effects on range of motion recovery in thumb stiff joint.

Methods and Findings

The aim of the first experiment was to examine the real-time effects of tetanic SES on the maximal volitional level of force over repeated contractions of the triceps brachii muscle. To address this goal, seventeen subjects participated voluntarily in this study. Two features of the muscular force were assessed: The peak force (1) and the impulse (2). These two dependent variables were measured during 500 sec - including 50 maximal force productions of 4 sec each- in two randomized conditions of VOL and SES. When considering the 50 trials as a whole, exerted force was higher in the SES than in the VOL condition for both peak force and impulse (P<.05). Over time, peak force and impulse decreased consistently in VOL starting between the 20th and 30th trials whereas they were maintained in SES condition (P<.05).

The aim of the second experiment was to compare the effects of VOL and SES on the range of flexion recovery of the stiff metacarpophalangeal joint following operative repair of the ulnar collateral ligament of the thumb. To address this goal, eight patients participated voluntarily. Range of motion, oedema and pain were assessed before and after the two randomised conditions of VOL and SES.

ELIGIBILITY:
Inclusion Criteria:

* loss of range of flexion in the involved metacarpophalangeal joint of at least ten degrees when compared to the opposite thumb
* more than eight weeks post-surgery

Exclusion Criteria:

* do not meet the inclusion criteria

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hand physical therapy center
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
range of motion | 1sec after joint mobilization
  Active range of motion was measured using a finger goniometer

SECONDARY OUTCOMES:
muscle force | During the muscle contraction
  The peak force and the impulse were measured during 500 sec in two randomized conditions of voluntary muscle contraction and electrically induced muscle contraction

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Nougier, PhD, Study Director — Université Joseph Fourier - TIMC IMAG laboratory
Locations (1):
- Université Joseph Fourier - TIMC IMAG laboratory, La Tronche, France

REFERENCES:
- [Background] Bostock S, Morris MA. The range of motion of the MP joint of the thumb following operative repair of the ulnar collateral ligament. J Hand Surg Br. 1993 Dec;18(6):710-1. doi: 10.1016/0266-7681(93)90227-7. PMID 8308425